CLINICAL TRIAL: NCT01101633
Title: The Effect of Sodium Alginate Containing Beverage on Appetite and Body Weight Regulation
Brief Title: The Effect of Sodium Alginate on Appetite Sensation
Acronym: B247Algobes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: SBiotek (Unknown)
Responsible Party: Arne Astrup, Prof. Dr. Med., Department of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-C-2008-088
Record Dates: First submitted 2009-08-25; First posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2009-08

CONDITIONS: Obesity; Overweight
Keywords: Appetite; Energy intake; gastric emptying; well being; Body weight
MeSH Terms: conditions — Obesity; Overweight; Body Weight | interventions — Alginates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 500 ml beverage containing alginate (3%)
  Interventions: Dietary Supplement: Alginate
- 2 (Active Comparator): 330 ml beverage containing alginate (3%)
  Interventions: Dietary Supplement: Alginate
- 3 (Placebo Comparator): 500 ml beverage without alginate (placebo)
  Interventions: Dietary Supplement: Placebo
- 4 (Placebo Comparator): 330 ml beverage without alginate (placebo)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alginate — a 500 ml alginate beverage per meal test
  Arms: 1
Dietary Supplement: Alginate — a 330 ml alginate beverage per meal test
  Arms: 2
Dietary Supplement: Placebo — a 500 ml placebo beverage per meal test
  Arms: 3
Dietary Supplement: Placebo — a 330 ml placebo beverage per meal test
  Arms: 4

SUMMARY:
The aim of the study is to investigate the effects of a low-calorie alginate containing fruit flavored beverage on appetite and body weight development.

DETAILED DESCRIPTION:
The project consists of two different studies:

Study I: A randomised controled meal test study aimed at studying the acute effect of the alginate-containing beverage on appetite sensation and spontaneous calorie intake (and safety i.e. nausea, well-being etc) in normal to overweight healthy subjects. Here, a placebo beverage or the alginate-containing beverage will be administered as a pre-load before a standardised breakfast meal. Subjective appetite sensation will be measured with Visual Analogue Scale (VAS) every 30 minutes four up to 5 hours. An additional beverage will be administered prior to an ad libitum lunch meal, where spontaneous water and energy intake will be registered.

Study II: Secondly the aim is to study the effects of a daily intake of a placebo or alginate-containing beverage on body weight and composition in a randomised parallel intervention study of 12 weeks duration. A total of app. 50 obese healthy adults will receive a hypocaloric diet and be randomised to consume either placebo or alginate-containing beverage before each of the three main meals every day. The development in body weight and composition and blood pressure will be monitored and blood samples will be analysed for markers related to the risk of CVD and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Normal to slight overweight (BMI: 22-28 kg/m2)
* 20-45 years of age

Exclusion Criteria:

* Smoking
* Daily medicine use (oral contraceptives excluded)
* Use of dietary supplements
* Blood donation 3 months prior to the study
* Hb<7.5 mmol/l
* Chronic illnesses such as hyperlipidemia, diabetes and inflammatory diseases
* Pregnancy or breastfeeding
* Elite athletes (>10 hours hard exercise/week)
* Vegetarians

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
appetite sensation | 5 hours

SECONDARY OUTCOMES:
Plasma insulin and glucose level | 5 hours
Well being and adverse events | 5 hours
gastric emptying | 5 hours
spontaneous calorie intake | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Dr. Med, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Human Nutrtion, University of Copenhagen, Frederiksberg, Copenhagen, Denmark

REFERENCES:
- [Derived] Georg Jensen M, Kristensen M, Belza A, Knudsen JC, Astrup A. Acute effect of alginate-based preload on satiety feelings, energy intake, and gastric emptying rate in healthy subjects. Obesity (Silver Spring). 2012 Sep;20(9):1851-8. doi: 10.1038/oby.2011.232. Epub 2011 Jul 21. PMID 21779093